CLINICAL TRIAL: NCT05967676
Title: Turkish Adaptation, Validity and Reliability of the Psychological Readiness of Injured Athlete to Return to Sport (PRIA-RS) Questionnaire
Brief Title: Psychological Readiness of Injured Athlete to Return to Sport
Acronym: PRIA-RS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, Lecturer, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16.12.2022
Record Dates: First submitted 2023-07-22; First posted 2023-08-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Athletic Injuries
Keywords: Validity; Reliability; Turkish Adaptation; Psychological Readiness; sports injury
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Adaptation, validity and reliability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (Experimental): athletes who have suffered a sports injury
  Interventions: Diagnostic Test: Turkish adaptation, validity and reliability

INTERVENTIONS:
Diagnostic Test: Turkish adaptation, validity and reliability — This study was conducted as "test-retest" design and the psychometric properties of PRIA-RS were examined in injured athletes

SUMMARY:
Clinicians are recommended to assess athletes during the rehabilitation phase to identify athletes with potentially maladaptive psychological responses to injury. Therefore, the Psychological Readiness of Injured Athlete to Return to Sport (PRIA-RS) questionnaire was developed to assess the athlete's psychological readiness to return to sport. The aim of this study was to adapt the PRIA-RS questionnaire into Turkish and to establish its validity and reliability. Serial approach method will be used while translating the questionnaire into Turkish. In order to evaluate the validity of PRIA-RS, The Re-injury Anxiety Inventory and Tampa Kinesiophobia Scale will be applied to the participants.

ELIGIBILITY:
Inclusion Criteria:

* athletes who have missed at least 2 months of training due to injury
* having an upper, lower extremity or spine injury

Exclusion Criteria:

* having a psychological disorder
* regular use of psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Psychological Readiness of Injured Athlete to Return to Sport (PRIA-RS) | Baseline
  The PRIA-RS questionnaire provides a comprehensive screening of psychological readiness for return to sport based on athlete-reported confidence, self-perception, insecurity and fear of re-injury at the end of competition. The PRIA-RS questionnaire consists of 10 questions with each question scored on a 5-point Likert scale (50 points total), with a higher score representing a more positive psychological response.
Re-injury Anxiety Inventory (RAI): | Baseline
  The questionnaire developed by Walker et al. to measure re-injury anxiety is a 4-point Likert-type questionnaire and consists of 28 items in total. The questionnaire consists of two subgroups including re-injury anxiety/concern about rehabilitation and re-injury anxiety/concern about return to sport and training. A higher score represents more re-injury anxiety.
Tampa kinesiophobia scale (TKS) | Baseline
  It is a 17-question scale developed to measure fear of movement/reinjury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. The scale uses a 4-point Likert scale (Strongly disagree=1, Strongly agree=4). A higher score represents more kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirtas G, Yilmaz Ozal S, Guzel NA. Cross-cultural adaptation, validation, and reliability testing of the psychological readiness of injured athlete to return to sport (PRIA-RS) questionnaire in Turkish athletes. J Bodyw Mov Ther. 2025 Oct;44:155-160. doi: 10.1016/j.jbmt.2025.05.034. Epub 2025 May 21. PMID 40954576